CLINICAL TRIAL: NCT03803904
Title: Graded Intensity Aerobic Exercise to Improve Cerebrovascular Function and Performance in Aged Veterans
Brief Title: Aerobic Exercise and Cerebrovascular Function
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: E2825-R
Record Dates: First submitted 2019-01-09; First posted 2019-01-15 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Aging
Keywords: exercise; brain health
MeSH Terms: conditions — Motor Activity | interventions — spindlin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Spin (Experimental): The intervention will take place three times a week for 12 weeks and will be led by a qualified instructor (an Exercise Physiologist with five years of experience conducting the intervention). The duration of each session will be increased by 1-2 minutes to a maximum time of 45 minutes per session based on the progression of the participants and the recommendation of the instructor. Because participants are initially sedentary and detrained, exercise intensity will begin at low levels (50% of maximal heart rate reserve, HRR) but will be increased by 5% every week (if deemed necessary by the instructor) to a maximum of 75% maximal HRR.
  Interventions: Other: Spin
- Control (Active Comparator): Participants in the control group will be equalized (frequency and duration) to the Spin group for contact and monitoring. As such they will report to the same facility and interact with the same experienced interventionist; however instead of progressive Spin exercise they will participate in sessions focused on balance and stretching. Similar to the aerobic intervention, these exercises will take place in a group setting and heart rate will be consistently monitored during each session to verify heart rate does not reach 50% HRR.
  Interventions: Other: Spin

INTERVENTIONS:
Other: Spin — The intervention will take place three times a week for 12 weeks and will be led by a qualified instructor (an Exercise Physiologist with five years of experience conducting the intervention). The duration of each session will be increased by 1-2 minutes to a maximum time of 45 minutes per session based on the progression of the participants and the recommendation of the instructor. Because participants are initially sedentary and detrained, exercise intensity will begin at low levels (50% of maximal heart rate reserve, HRR) but will be increased by 5% every week (if deemed necessary by the instructor) to a maximum of 75% maximal HRR.

SUMMARY:
This proposal will evaluate two brain health measures, cerebrovascular perfusion and cerebrovascular reactivity (CVR), before and after a proven, interval-based, aerobic exercise intervention in older Veterans. The hypothesis is that the 12-week aerobic exercise intervention (Spin) will increase perfusion and improve CVR in brain regions susceptible to age-related decline. This information will inform the impact of exercise on cerebrovascular health which is known to be negatively impacted in aging and implicated in the development of neurogenerative disease. This information will also aid the investigators' continued efforts of clinical implementation of evidence-based exercise interventions in the local Atlanta VA and surround region.

DETAILED DESCRIPTION:
To address the growing healthcare challenges of an aging Veteran population it is critical to understand effective rehabilitation techniques that mitigate age-related co-morbidity and improve quality of life. To date, exercise is one of a few proven interventions that attenuates age-related declines in brain health and function. A consistent but unexplained finding in many of these studies is a change in the cortical activation pattern during task, assessed using blood-oxygen-level dependent (BOLD) signal with fMRI that corresponds with improved task performance. Two key metrics of cerebrovascular health and functioning that are underexplored but may influence the documented changes in the BOLD response that is observed with post-aerobic activity are: 1) changes in resting or basal cerebral blood flow (perfusion) to key brain regions; and 2) changes in the ability of cerebrovasculature to dilate in the face of increased demand, termed cerebrovascular reactivity (CVR). The investigators' goal is to quantify the impact of aerobic exercise on cerebrovascular function and how both perfusion and CVR contributes to the BOLD signal during task-based fMRI. Consistent with the investigators' previous aging and exercise studies participants will complete one of two conditions; 1) an aerobic, interval-training intervention (Spin; n= 44), or 2) a non-aerobic, stretching control condition (Control; n=44). Cardiovascular fitness, arterial spin labeling for basal cerebral perfusion, CVR, task-based fMRI (cognitive-executive and motor), and behavioral outcomes will be assessed before and after the interventions. The specific aims will determine the effect of a 12-week aerobic exercise intervention on changes in cerebral perfusion and CVR in older Veterans. The investigators hypothesize that compared to the Control group, the aerobically-trained group will have increased basal perfusion and CVR in areas that demonstrate age-related decline and that have been demonstrated to be malleable to aerobic exercise (inferior frontal and motor cortices).

Research over the last few decades have driven the continual promotion of exercise as one of the most impactful interventions of central nervous system health and function. At the forefront of much of this research is the use of task-based fMRI BOLD to quantify beneficial changes in cortical function following aerobic exercise. While transformative, the true impact of this research is limited in scope until the investigators can define the influence of cerebrovascular function on the well-documented beneficial change in BOLD response. The investigators do know that older adults who are physically active have improved vascular health but do not know the full impact of an exercise intervention on cerebrovascular health. If the hypotheses of improved perfusion and CVR is supported it would inform current intervention strategies and would add important additional information about the potential of exercise to improve brain health in aging. This would have implications for aging Veterans at risk for neurodegenerative disease brought on by cerebrovascular dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 65-80 who do not regularly exercise

  * defined as exercising less than 20 minutes twice per week
* Are willing and able to cooperate with assessments and interventions
* Participant will be quantified at or below the "poor" range for cardiovascular fitness as assessed by a volume of oxygen (VO2) test

  * 26.0 ml/kg/min for males
  * 21.0 ml/kg/min for females)
* 26 on the MoCA to meet the criteria for cognitively intact
* Participants will be free from diseases affecting cognition or that would interfere with their ability to engage in aerobic exercise - including but not limited to:

  * chronic heart
  * liver
  * kidney disease
* Free from diseases/injuries directly affecting brain functions - including but not limited to:

  * significant closed head injury
  * open intracranial wounds
  * stroke
  * epilepsy
  * degenerative diseases of the nervous system
* All subjects will speak English as a primary language and will have at minimum a high school diploma so that behavioral/cognitive measures reflect effects of aging and aerobic exercise and not unfamiliarity with the English language or a lack of education

Exclusion Criteria:

* Potential participants with major psychiatric disorder - including but not limited to:

  * psychosis
  * major depression
  * bipolar disorder
* Individuals with ongoing drug or alcohol abuse and severe hypertension (systolic BP > 200 or diastolic BP > 110 mm Hg or subjects taking three or more antihypertensive medications
* Participants must not have conditions incompatible with MRI - including but not limited to:

  * ferrous metal implants
  * cardiac pacemakers or similar devices
  * claustrophobia
  * morbid obesity
* Persons engaging in significant skilled manual movements regularly will be excluded so that behavioral/motor measures reflect the effects of age and aerobic exercise and not the effects of frequent practice

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2025-01-10 (Actual); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Arterial Spin Labeling (ASL) to Measure Cerebral Blood Flow Change | At the Pre-intervention assessment and 12-weeks following at the Post intervention assessment
  ASL is a robust, sensitive and specific, non-invasive technique used for determining the amount of arterial blood flow to the whole brain or a particular ROI.47,48 In ASL, arterial blood water is magnetically labeled at the ROI by applying a 180 degree radiofrequency inversion pulse, resulting in magnetization of the blood water. The labeled water exchanges with tissue water, which alters the tissue magnetization and the image intensity creating a "tag" image. This process is repeated without magnetically labeling the arterial blood water, thus creating a "control" image. Subtracting the control and tag images produces the perfusion imaging which reflects the amount of arterial blood delivered to each voxel within the region of interest, termed difference signal.

SECONDARY OUTCOMES:
Cerebrovascular reactivity (CVR) using a hypercapnic CO2 response test change | At the Pre-intervention assessment and 12-weeks following at the Post intervention assessment
  CVR will be assessed using 5% CO2 challenge while continuously acquiring MR images. This method has been extensively used and is the most suitable vasoactive stimulus.33,34 Briefly, the CO2 air (5% CO2, 21% O2 and 74% N2) will be administered via an air bag with a valve to switch between room air and CO2 air in the bag. A mouth piece and a nose clip will be used to achieve mouth-only breathing. A research staff member will be inside the magnet room throughout the experiment to switch the valve and to monitor the subject. Physiologic parameters, including end-tidal (Et) CO2 and breathing rate will be monitored and recorded during the experiments.

CONTACTS AND LOCATIONS:
Overall Officials: Joe R. Nocera, PhD, Principal Investigator — Atlanta VA Medical and Rehab Center, Decatur, GA
Locations (1):
- Atlanta VA Medical and Rehab Center, Decatur, GA, Decatur, Georgia, United States

IPD SHARING:
Plan to Share IPD: No